# **Study Information Sheet for Patients**

Study Title: A pilot study to test the acceptability and feasibility of a brief discussion to help

patients formulate their goals for medical care in the emergency department

Version: 5/3/2018

Principal Investigator (PI): Kei Ouchi, MD, MPH

NCT03208530

Version 2018-05-03 

**Purpose of the Research:** We want to help advance care planning (ACP) discussions for older adults with serious illness in the emergency department (ED).

Funder of the Research: Emergency Medicine Foundation and National Institute on Aging

How we obtained your name and contact information: We asked your Brigham and

Women's Hospital ED clinicians to identify you.

#### Why are we asking you to participate?

We are asking you to participate because we want to understand what would help patients like you to talk to your outpatient doctors about advance care planning.

## How many people are anticipated to participate?

We are asking about 125 patients to take part in this study.

## How long it will take to complete the study and what does it entail?

The study will take place in the Emergency Department (including the ED observation unit). In order to confirm that you are qualified for the study, we will perform two short tests before the interview. If you are qualified, we will ask you to complete some survey questions and then study clinicians will conduct a brief motivational interview with you. We anticipate that this will take about 10-20 minutes. After the encounter, we may also interview you for 10 to 15 minutes to ask you about how you felt about it. With your permission, we will video-record your motivational interview with the study clinician, as well as the interview to understand how you felt about the interaction to make sure we understand you correctly. We will also contact you in about seven days and one month after the interview to ask you some survey questions. These surveys can be completed in about 10 minutes: i. over the phone (we will schedule for the specific time of your convenience); or ii. by mail mailed survey with a return postage; or iii. inperson by a research assistant at the next doctor's appointment, whichever you prefer (we will find out when that appointment will be from you or using your medical records). If you choose to complete the surveys by mail, we will provide you with return postage and place a call to remind you when to complete them. If you choose to complete the surveys over the phone, with your permission, we will make a voice recording of the conversation, which will be stored on a secure drive. We will plan to continue enrollment until we complete 125 doctor-patient encounters total.

**Payment:** For participation in this study, you will receive a certificate of participation and a compensation of \$5 for completing the motivational interview in the ED. In addition, we will send a "Thank You" postcard (see attached) and a total of \$10 to all participants at the time of outcome survey (the total compensation of the entire study is \$15).

Version 2018-05-03 

## **Confidentiality and Data Security**

Your information and responses will be de-identified (we will not be able to match specific data to specific participant). Study information will be stored in a secure location. Only the study staff can review your study information.

## What are the risks associated with participation?

There is no clear foreseeable risk associated with participation in this study other than 30 to 35 extra minutes of your time during your stay in the ED or ED observation unit and during the follow-up phone calls. We will ask you to think about your illness and care goals in the future, which may make you anxious. We can help you deal with these feelings if needed. Your participation is voluntary and you may stop at any time. Deciding not to participate will have no effect on your care.

#### **Questions:**

The PI can be contacted at the following 24 hours / day and 7 days per week:

Cell - 857-205-4947

Email - kouchi@partners.org

If you'd like to speak to someone not involved in this research about your rights as a research subject, or any concerns or complaints you may have about the research, contact the Partners Human Research Committee at 857-282-1900.

Version 2018-05-03 